CLINICAL TRIAL: NCT03314922
Title: A Phase 1b, Open-Label, Dose-Escalation Study for the Safety, Tolerability, and Pharmacokinetics of INCB050465 in Japanese Subjects With Previously Treated B-Cell Lymphoma (CITADEL-111)
Brief Title: A Study of INCB050465 in Japanese Subjects With Previously Treated B-Cell Lymphoma (CITADEL-111)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-111/CITADEL-111; Parsaclisib (Other: Incyte Corporation)
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma
Keywords: Diffuse large B-cell lymphoma (DLBCL); follicular lymphoma (FL); marginal zone lymphoma (MZL); mantle cell lymphoma (MCL); phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Parsaclisib (Experimental)
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib administered orally once daily for 8 weeks at the protocol-defined dose, followed by a once-weekly regimen at the same dose.
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of parsaclisib in the treatment of Japanese participants diagnosed with previously-treated B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* First generation Japanese; subject was born in Japan and has not lived outside of Japan for > 10 years, and subject can trace maternal and paternal Japanese ancestry.
* Histologically confirmed aggressive/indolent DLBCL, FL, MZL, or MCL.
* Previously received at least 1 prior line of systemic therapy with documented progression, and there is no further effective standard anticancer therapy available.
* Willing to undergo an incisional or excisional lymph node or tissue biopsy or to provide a lymph node or tissue biopsy from the most recent available archival tissue.
* Life expectancy > 3 months.
* Eastern Cooperative Oncology Group performance status of 0 to 2.
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Evidence of transformed non-Hodgkin's lymphoma histologies.
* Histologically confirmed, rare non-Hodgkin's B-cell subtypes.
* History of central nervous system lymphoma (either primary or metastatic) or leptomeningeal disease.
* Prior treatment with idelalisib, other selective PI3Kδ inhibitors, or a pan-phosphatidylinositol 3 kinase (PI3K) inhibitor.
* Allogeneic stem cell transplant within the last 6 months or autologous stem cell transplant within the last 3 months before the date of the first dose of study drug.
* Active graft-versus-host disease.
* History of stroke or intracranial hemorrhage within 6 months of study drug administration.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment or exposure to a live vaccine within 30 days of the date of the first dose of study drug.
* Known human immunodeficiency virus infection.
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to approximately 1 year
  TEAE defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Changes in pharmacodynamic (PD) markers of B-cell activation in plasma | Up to 24 weeks
  Markers of B-cell activation (eg, B-cell activating factor, interleukin-10, B-cell attracting chemokine) and other plasma analytes will be analyzed for correlation with safety and clinical outcome.
Objective response rate | Up to approximately 1 year
  Defined as the percentage of subjects with complete response (CR)/complete metabolic response (CMR) and partial response (PR)/ partial metabolic response (PMR), as determined by investigator assessment of response according to response criteria for lymphomas.
Duration of response | Up to approximately 1 year
  Defined as the time from first documented evidence of CR/CMR or PR/PMR until disease progression or death from any cause among subjects who achieve an objective response.
Progression-free survival | Up to approximately 1 year
  Defined as the time from the date of the first dose of study drug until the earliest date of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Cinthya Coronado, MD, Study Director — Incyte Corporation
Locations (6):
- Japan (6):
  - Aichi Cancer Center Hospital, Aichi
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Cancer Institute Hospital of Jfcr, Kōtoku
  - Nagoya City University Hospital, Nagoya
  - Tohoku University Hospital, Sendai
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available at the end of trial or termination of trial. The following data will be made available: safety, PK and PD, efficacy, and subject characteristics. The results of the trial will be published. In addition, data as documented in study CSR will be made available upon request.